CLINICAL TRIAL: NCT00975195
Title: A Randomised, Double-blind, Active-controlled Study to Evaluate the Impact of Stepwise Withdrawal of Inhaled Corticosteroid Treatment in Patients With Severe to Very Severe Chronic Obstructive Pulmonary Disease (COPD) on Optimized Bronchodilator Therapy
Brief Title: Inhaled Corticosteroid Withdrawal in Patients With Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 352.2046; 2007-002522-29 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- fluticasone high dose (Experimental): fluticasone priopionate high dose and tiotropium inhalation and salmeterol xinafoate
  Interventions: Drug: tiotropium inhalation; Drug: salmeterol xinafoate; Drug: fluticasone propionate
- fluticasone medium & low doses (Experimental): fluticasone priopionate medium and high doses; and tiotropium inhalation; and salmeterol xinafoate; and placebo matched to fluticasone priopionate
  Interventions: Drug: tiotropium inhalation; Drug: salmeterol xinafoate; Drug: fluticasone propionate; Drug: placebo matched for fluticasone propionate

INTERVENTIONS:
Drug: tiotropium inhalation
Drug: salmeterol xinafoate
Drug: fluticasone propionate
Drug: placebo matched for fluticasone propionate
  Arms: fluticasone medium & low doses

SUMMARY:
This is a randomised study to be conducted in patients with severe to very severe Chronic Obstructive Pulmonary Disease (COPD) to establish whether there is a need for these patients to be continuously treated with an inhaled corticosteroid on top of two potent long-acting bronchodilators. The study also aims to identify the type of patients who are likely to benefit from inhaled corticosteroid maintenance therapy.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged 40 years or more
2. Severe to very severe chronic obstructive pulmonary disease (COPD)
3. Current or ex-smoker with smoking history of at least 10 pack years
4. At least one documented exacerbation of COPD in previous year

Exclusion criteria:

1. Significant diseases other than COPD; significant alcohol or drug abuse
2. Current clinical diagnosis of asthma requiring steroid treatment
3. History of thoracotomy with pulmonary resection
4. Regular use of daytime oxygen
5. Recent history (within 3 months) of myocardial infarction
6. Recent (within 6 weeks) respiratory infection or COPD exacerbation
7. Recent (within 6 weeks) treatment with systemic corticosteroids at doses in excess of 5milligram / day
8. Recent (within 3 months) unstable or life-threatening cardiac arrhythmia requiring intervention
9. Recent (within 1 year) hospitalisation for cardiac failure
10. Malignancy requiring chemotherapy or radiotherapy
11. Clinical diagnosis of bronchiectasis
12. Pregnant or nursing women
13. Known hypersensitivity to study drugs
14. Current or recent (within 30 days) participation in another clinical study
15. Current participation in or recent completion (within 4 weeks) of a pulmonary rehabilitation program

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2488 (Actual)
Dates: Start 2009-02; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (222):
- Australia (6):
  - 352.2046.61006 Boehringer Ingelheim Investigational Site, Concord, New South Wales
  - 352.2046.61001 Boehringer Ingelheim Investigational Site, Glebe, New South Wales
  - 352.2046.61002 Boehringer Ingelheim Investigational Site, Westmead, New South Wales
  - 352.2046.61004 Boehringer Ingelheim Investigational Site, Daw Park, South Australia
  - 352.2046.61003 Boehringer Ingelheim Investigational Site, Toorak Gardens, South Australia
  - 352.2046.61005 Boehringer Ingelheim Investigational Site, Woodville, South Australia
- Belgium (11):
  - 352.2046.32002 Boehringer Ingelheim Investigational Site, Brussels
  - 352.2046.32016 Boehringer Ingelheim Investigational Site, Brussels
  - 352.2046.32015 Boehringer Ingelheim Investigational Site, Eupen
  - 352.2046.32017 Boehringer Ingelheim Investigational Site, Gilly
  - 352.2046.32014 Boehringer Ingelheim Investigational Site, Herentals
  - 352.2046.32006 Boehringer Ingelheim Investigational Site, Jambes
  - 352.2046.32008 Boehringer Ingelheim Investigational Site, Lebbeke
  - 352.2046.32001 Boehringer Ingelheim Investigational Site, Leuven
  - 352.2046.32004 Boehringer Ingelheim Investigational Site, Middelheim
  - 352.2046.32010 Boehringer Ingelheim Investigational Site, Montigny-le-Tilleul
  - 352.2046.32013 Boehringer Ingelheim Investigational Site, Turnhout
- Brazil (5):
  - 352.2046.55002 Boehringer Ingelheim Investigational Site, Goiânia
  - 352.2046.55005 Boehringer Ingelheim Investigational Site, Goiânia
  - 352.2046.55001 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 352.2046.55006 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 352.2046.55003 Boehringer Ingelheim Investigational Site, São Paulo
- Bulgaria (8):
  - 352.2046.35905 Boehringer Ingelheim Investigational Site, Burgas
  - 352.2046.35902 Boehringer Ingelheim Investigational Site, Rousse
  - 352.2046.35904 Boehringer Ingelheim Investigational Site, Sofia
  - 352.2046.35906 Boehringer Ingelheim Investigational Site, Sofia
  - 352.2046.35907 Boehringer Ingelheim Investigational Site, Sofia
  - 352.2046.35908 Boehringer Ingelheim Investigational Site, Sofia
  - 352.2046.35903 Boehringer Ingelheim Investigational Site, Stara Zagora
  - 352.2046.35909 Boehringer Ingelheim Investigational Site, Veliko Tarnovo
- China (8):
  - 352.2046.86002 Boehringer Ingelheim Investigational Site, Beijing
  - 352.2046.86003 Boehringer Ingelheim Investigational Site, Beijing
  - 352.2046.86006 Boehringer Ingelheim Investigational Site, Beijing
  - 352.2046.86008 Boehringer Ingelheim Investigational Site, Chongqing
  - 352.2046.86001 Boehringer Ingelheim Investigational Site, Guangzhou
  - 352.2046.86004 Boehringer Ingelheim Investigational Site, Shanghai
  - 352.2046.86005 Boehringer Ingelheim Investigational Site, Shanghai
  - 352.2046.86007 Boehringer Ingelheim Investigational Site, Wuhan
- Denmark (3):
  - 352.2046.45001 Boehringer Ingelheim Investigational Site, Aarhus C
  - 352.2046.45003 Boehringer Ingelheim Investigational Site, København NV
  - 352.2046.45002 Boehringer Ingelheim Investigational Site, Odense C
- France (33):
  - 352.2046.3317A Boehringer Ingelheim Investigational Site, Brest
  - 352.2046.3317B Boehringer Ingelheim Investigational Site, Brest
  - 352.2046.3317C Boehringer Ingelheim Investigational Site, Brest
  - 352.2046.3320A Boehringer Ingelheim Investigational Site, Castelnau-le-Lez
  - 352.2046.3320B Boehringer Ingelheim Investigational Site, Castelnau-le-Lez
  - 352.2046.3320C Boehringer Ingelheim Investigational Site, Castelnau-le-Lez
  - 352.2046.3335A Boehringer Ingelheim Investigational Site, Clermont-Ferrand
  - 352.2046.3314A Boehringer Ingelheim Investigational Site, Forbach
  - 352.2046.3301A Boehringer Ingelheim Investigational Site, Marseille
  - 352.2046.3333A Boehringer Ingelheim Investigational Site, Marseille
  - 352.2046.3326A Boehringer Ingelheim Investigational Site, Montpellier
  - 352.2046.3326C Boehringer Ingelheim Investigational Site, Montpellier
  - 352.2046.3325A Boehringer Ingelheim Investigational Site, Nantes
  - 352.2046.3325C Boehringer Ingelheim Investigational Site, Nantes
  - 352.2046.3325D Boehringer Ingelheim Investigational Site, Nantes
  - 352.2046.3334A Boehringer Ingelheim Investigational Site, Nantes
  - 352.2046.3324A Boehringer Ingelheim Investigational Site, Nîmes
  - 352.2046.3332A Boehringer Ingelheim Investigational Site, Nîmes
  - 352.2046.3332B Boehringer Ingelheim Investigational Site, Nîmes
  - 352.2046.3332C Boehringer Ingelheim Investigational Site, Nîmes
  - 352.2046.3331A Boehringer Ingelheim Investigational Site, Perpignan
  - 352.2046.3331B Boehringer Ingelheim Investigational Site, Perpignan
  - 352.2046.3331C Boehringer Ingelheim Investigational Site, Perpignan
  - 352.2046.3329A Boehringer Ingelheim Investigational Site, Saint-Laurent-du-Var
  - 352.2046.3329B Boehringer Ingelheim Investigational Site, Saint-Laurent-du-Var
  - 352.2046.3302A Boehringer Ingelheim Investigational Site, Saint-Pierre
  - 352.2046.3302B Boehringer Ingelheim Investigational Site, Saint-Pierre
  - 352.2046.3302C Boehringer Ingelheim Investigational Site, Saint-Pierre
  - 352.2046.3302D Boehringer Ingelheim Investigational Site, Saint-Pierre
  - 352.2046.3336A Boehringer Ingelheim Investigational Site, Toulouse
  - 352.2046.3336B Boehringer Ingelheim Investigational Site, Toulouse
  - 352.2046.3336C Boehringer Ingelheim Investigational Site, Toulouse
  - 352.2046.3337A Boehringer Ingelheim Investigational Site, Toulouse
- Germany (19):
  - 352.2046.49012 Boehringer Ingelheim Investigational Site, Berlin
  - 352.2046.49020 Boehringer Ingelheim Investigational Site, Berlin
  - 352.2046.49021 Boehringer Ingelheim Investigational Site, Berlin
  - 352.2046.49008 Boehringer Ingelheim Investigational Site, Bochum
  - 352.2046.49003 Boehringer Ingelheim Investigational Site, Cologne
  - 352.2046.49019 Boehringer Ingelheim Investigational Site, Cottbus
  - 352.2046.49002 Boehringer Ingelheim Investigational Site, Donaustauf
  - 352.2046.49013 Boehringer Ingelheim Investigational Site, Frankfurt
  - 352.2046.49025 Boehringer Ingelheim Investigational Site, Frankfurt
  - 352.2046.49023 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 352.2046.49024 Boehringer Ingelheim Investigational Site, Geesthacht
  - 352.2046.49022 Boehringer Ingelheim Investigational Site, Gelnhausen
  - 352.2046.49001 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 352.2046.49006 Boehringer Ingelheim Investigational Site, Heidelberg
  - 352.2046.49014 Boehringer Ingelheim Investigational Site, Immenhausen
  - 352.2046.49016 Boehringer Ingelheim Investigational Site, Kiel
  - 352.2046.49004 Boehringer Ingelheim Investigational Site, Mainz
  - 352.2046.49005 Boehringer Ingelheim Investigational Site, Marburg
  - 352.2046.49015 Boehringer Ingelheim Investigational Site, München
- Greece (11):
  - 352.2046.30003 Boehringer Ingelheim Investigational Site, Athens
  - 352.2046.30004 Boehringer Ingelheim Investigational Site, Athens
  - 352.2046.30005 Boehringer Ingelheim Investigational Site, Athens
  - 352.2046.30007 Boehringer Ingelheim Investigational Site, Athens
  - 352.2046.30008 Boehringer Ingelheim Investigational Site, Athens
  - 352.2046.30011 Boehringer Ingelheim Investigational Site, Athens
  - 352.2046.30012 Boehringer Ingelheim Investigational Site, Athens
  - 352.2046.30006 Boehringer Ingelheim Investigational Site, Heraklion
  - 352.2046.30009 Boehringer Ingelheim Investigational Site, Larissa
  - 352.2046.30001 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 352.2046.30002 Boehringer Ingelheim Investigational Site, Thessaloniki
- Hungary (7):
  - 352.2046.36003 Boehringer Ingelheim Investigational Site, Cegléd
  - 352.2046.36002 Boehringer Ingelheim Investigational Site, Deszk
  - 352.2046.36004 Boehringer Ingelheim Investigational Site, Komárom
  - 352.2046.36006 Boehringer Ingelheim Investigational Site, Pécs
  - 352.2046.36001 Boehringer Ingelheim Investigational Site, Szarvas
  - 352.2046.36005 Boehringer Ingelheim Investigational Site, Százhalombatta
  - 352.2046.36011 Boehringer Ingelheim Investigational Site, Szigetszentmiklós
- Italy (8):
  - 352.2046.39002 Boehringer Ingelheim Investigational Site, Catania
  - 352.2046.39007 Boehringer Ingelheim Investigational Site, Cona
  - 352.2046.39005 Boehringer Ingelheim Investigational Site, Foggia
  - 352.2046.39003 Boehringer Ingelheim Investigational Site, Modena
  - 352.2046.39006 Boehringer Ingelheim Investigational Site, Montescano (pv)
  - 352.2046.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 352.2046.39004 Boehringer Ingelheim Investigational Site, Sesto S. Giovanni (mi)
  - 352.2046.39008 Boehringer Ingelheim Investigational Site, Tradate (va)
- Netherlands (4):
  - 352.2046.31004 Boehringer Ingelheim Investigational Site, Heerlen
  - 352.2046.31001 Boehringer Ingelheim Investigational Site, Leeuwarden
  - 352.2046.31003 Boehringer Ingelheim Investigational Site, Rotterdam
  - 352.2046.31002 Boehringer Ingelheim Investigational Site, Veldhoven
- New Zealand (7):
  - 352.2046.64007 Boehringer Ingelheim Investigational Site, Auckland NZ
  - 352.2046.64003 Boehringer Ingelheim Investigational Site, Christchurch
  - 352.2046.64004 Boehringer Ingelheim Investigational Site, Dunedin
  - 352.2046.64006 Boehringer Ingelheim Investigational Site, Hamilton
  - 352.2046.64001 Boehringer Ingelheim Investigational Site, Newtown Wellington NZ
  - 352.2046.64005 Boehringer Ingelheim Investigational Site, Otahuhu New Zealand
  - 352.2046.64002 Boehringer Ingelheim Investigational Site, Tauranga
- Philippines (8):
  - 352.2046.63001 Boehringer Ingelheim Investigational Site, Caloocan
  - 352.2046.63009 Boehringer Ingelheim Investigational Site, City of Muntinlupa
  - 352.2046.63003 Boehringer Ingelheim Investigational Site, Manila
  - 352.2046.63004 Boehringer Ingelheim Investigational Site, Manila
  - 352.2046.63005 Boehringer Ingelheim Investigational Site, Quezon
  - 352.2046.63007 Boehringer Ingelheim Investigational Site, Quezon
  - 352.2046.63006 Boehringer Ingelheim Investigational Site, Quezon City
  - 352.2046.63008 Boehringer Ingelheim Investigational Site, Quezon City
- Poland (8):
  - 352.2046.48006 Boehringer Ingelheim Investigational Site, Bytom
  - 352.2046.48003 Boehringer Ingelheim Investigational Site, Ostrow Wielkopolska
  - 352.2046.48001 Boehringer Ingelheim Investigational Site, Poznan
  - 352.2046.48002 Boehringer Ingelheim Investigational Site, Poznan
  - 352.2046.48009 Boehringer Ingelheim Investigational Site, Rzeszów
  - 352.2046.48011 Boehringer Ingelheim Investigational Site, Tarnowskie Góry
  - 352.2046.48005 Boehringer Ingelheim Investigational Site, Warsaw
  - 352.2046.48007 Boehringer Ingelheim Investigational Site, Wroclaw
- Russia (9):
  - 352.2046.07006 Boehringer Ingelheim Investigational Site, Ivanovo
  - 352.2046.07008 Boehringer Ingelheim Investigational Site, Moscow
  - 352.2046.07009 Boehringer Ingelheim Investigational Site, Moscow
  - 352.2046.07001 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 352.2046.07002 Boehringer Ingelheim Investigational Site, Samara
  - 352.2046.07003 Boehringer Ingelheim Investigational Site, Saratov
  - 352.2046.07004 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 352.2046.07005 Boehringer Ingelheim Investigational Site, Yaroslavl
  - 352.2046.07011 Boehringer Ingelheim Investigational Site, Yekaterinburg
- South Africa (7):
  - 352.2046.27002 Boehringer Ingelheim Investigational Site, Bellville
  - 352.2046.27001 Boehringer Ingelheim Investigational Site, Cape Town
  - 352.2046.27003 Boehringer Ingelheim Investigational Site, Cape Town
  - 352.2046.27006 Boehringer Ingelheim Investigational Site, eManzimtoti
  - 352.2046.27007 Boehringer Ingelheim Investigational Site, Pretoria
  - 352.2046.27005 Boehringer Ingelheim Investigational Site, Somerset West
  - 352.2046.27004 Boehringer Ingelheim Investigational Site, Tygerberg
- Spain (9):
  - 352.2046.34008 Boehringer Ingelheim Investigational Site, Badajoz
  - 352.2046.34002 Boehringer Ingelheim Investigational Site, Barakaldo (Bilbao)
  - 352.2046.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 352.2046.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 352.2046.34009 Boehringer Ingelheim Investigational Site, L'Hospitalet de Llobregat
  - 352.2046.34006 Boehringer Ingelheim Investigational Site, Palma de Mallorca
  - 352.2046.34010 Boehringer Ingelheim Investigational Site, Pozuelo de Alarcón
  - 352.2046.34013 Boehringer Ingelheim Investigational Site, Salt (Girona)
  - 352.2046.34011 Boehringer Ingelheim Investigational Site, Seville
- Taiwan (6):
  - 352.2046.88607 Boehringer Ingelheim Investigational Site, Dawan
  - 352.2046.88608 Boehringer Ingelheim Investigational Site, Dawan
  - 352.2046.88606 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 352.2046.88604 Boehringer Ingelheim Investigational Site, Taichung
  - 352.2046.88601 Boehringer Ingelheim Investigational Site, Taipei
  - 352.2046.88603 Boehringer Ingelheim Investigational Site, Taipei
- Tunisia (5):
  - 352.2046.2161A Boehringer Ingelheim Investigational Site, Aryanah
  - 352.2046.2162A Boehringer Ingelheim Investigational Site, Aryanah
  - 352.2046.2165A Boehringer Ingelheim Investigational Site, Sfax
  - 352.2046.2164A Boehringer Ingelheim Investigational Site, Sousse
  - 352.2046.2163A Boehringer Ingelheim Investigational Site, Tunis
- Turkey (Türkiye) (17):
  - 352.2046.90009 Boehringer Ingelheim Investigational Site, Ankara
  - 352.2046.90019 Boehringer Ingelheim Investigational Site, Ankara
  - 352.2046.90016 Boehringer Ingelheim Investigational Site, Bursa
  - 352.2046.90010 Boehringer Ingelheim Investigational Site, Denizli
  - 352.2046.90003 Boehringer Ingelheim Investigational Site, Istanbul
  - 352.2046.90004 Boehringer Ingelheim Investigational Site, Istanbul
  - 352.2046.90006 Boehringer Ingelheim Investigational Site, Istanbul
  - 352.2046.90008 Boehringer Ingelheim Investigational Site, Istanbul
  - 352.2046.90012 Boehringer Ingelheim Investigational Site, Istanbul
  - 352.2046.90017 Boehringer Ingelheim Investigational Site, Istanbul
  - 352.2046.90011 Boehringer Ingelheim Investigational Site, Izmir
  - 352.2046.90014 Boehringer Ingelheim Investigational Site, Izmir
  - 352.2046.90018 Boehringer Ingelheim Investigational Site, Izmir
  - 352.2046.90005 Boehringer Ingelheim Investigational Site, İzmit
  - 352.2046.90007 Boehringer Ingelheim Investigational Site, Kayseri
  - 352.2046.90001 Boehringer Ingelheim Investigational Site, Mersin
  - 352.2046.90002 Boehringer Ingelheim Investigational Site, Samsun
- Ukraine (7):
  - 352.2046.38007 Boehringer Ingelheim Investigational Site, Ivano-Frankivsk
  - 352.2046.38002 Boehringer Ingelheim Investigational Site, Kharkiv
  - 352.2046.38003 Boehringer Ingelheim Investigational Site, Kharkiv
  - 352.2046.38004 Boehringer Ingelheim Investigational Site, Kiev
  - 352.2046.38006 Boehringer Ingelheim Investigational Site, Kiev
  - 352.2046.38005 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 352.2046.38001 Boehringer Ingelheim Investigational Site, Vinnytsia
- United Kingdom (16):
  - 352.2046.44008 Boehringer Ingelheim Investigational Site, Baillieston, Glasgow
  - 352.2046.44009 Boehringer Ingelheim Investigational Site, Barnsley
  - 352.2046.44018 Boehringer Ingelheim Investigational Site, Belfast
  - 352.2046.44010 Boehringer Ingelheim Investigational Site, Birmingham
  - 352.2046.44003 Boehringer Ingelheim Investigational Site, Cambridge
  - 352.2046.44026 Boehringer Ingelheim Investigational Site, Chertsey
  - 352.2046.44006 Boehringer Ingelheim Investigational Site, Chesterfield
  - 352.2046.44012 Boehringer Ingelheim Investigational Site, Cottingham, Hull
  - 352.2046.44028 Boehringer Ingelheim Investigational Site, Inverness
  - 352.2046.44016 Boehringer Ingelheim Investigational Site, Isleworth
  - 352.2046.44002 Boehringer Ingelheim Investigational Site, Liverpool
  - 352.2046.44001 Boehringer Ingelheim Investigational Site, London
  - 352.2046.44017 Boehringer Ingelheim Investigational Site, Norwich
  - 352.2046.44021 Boehringer Ingelheim Investigational Site, Sheffield
  - 352.2046.44019 Boehringer Ingelheim Investigational Site, Sunderland
  - 352.2046.44025 Boehringer Ingelheim Investigational Site, Windsor

REFERENCES:
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Watz H, Tetzlaff K, Magnussen H, Mueller A, Rodriguez-Roisin R, Wouters EFM, Vogelmeier C, Calverley PMA. Spirometric changes during exacerbations of COPD: a post hoc analysis of the WISDOM trial. Respir Res. 2018 Dec 13;19(1):251. doi: 10.1186/s12931-018-0944-3. PMID 30545350
- [Derived] Watz H, Tetzlaff K, Wouters EF, Kirsten A, Magnussen H, Rodriguez-Roisin R, Vogelmeier C, Fabbri LM, Chanez P, Dahl R, Disse B, Finnigan H, Calverley PM. Blood eosinophil count and exacerbations in severe chronic obstructive pulmonary disease after withdrawal of inhaled corticosteroids: a post-hoc analysis of the WISDOM trial. Lancet Respir Med. 2016 May;4(5):390-8. doi: 10.1016/S2213-2600(16)00100-4. Epub 2016 Apr 7. PMID 27066739
- [Derived] Magnussen H, Disse B, Rodriguez-Roisin R, Kirsten A, Watz H, Tetzlaff K, Towse L, Finnigan H, Dahl R, Decramer M, Chanez P, Wouters EF, Calverley PM; WISDOM Investigators. Withdrawal of inhaled glucocorticoids and exacerbations of COPD. N Engl J Med. 2014 Oct 2;371(14):1285-94. doi: 10.1056/NEJMoa1407154. Epub 2014 Sep 8. PMID 25196117

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluticasone Maintenance: 18μg tiotropium administered by oral inhalation once daily (q.d.), 50μg salmeterol and 500μg fluticasone, each administered by oral inhalation twice daily (b.i.d) for 6 weeks (open-label run in period), followed by 18 μg tiotropium q.d., 50 μg salmeterol b.i.d.,and 500 μg fluticasone b.i.d. for 52 weeks (randomised treatment period).
- Fluticasone Withdrawal: 18μg tiotropium administered by oral inhalation once daily (q.d.), 50μg salmeterol and 500μg fluticasone, each administered by oral inhalation twice daily (b.i.d) for 6 weeks (open-label run in period), followed by 18 μg tiotropium q.d.and 50 μg salmeterol b.i.d. for 52 weeks, in combination with a stepwise withdrawal of fluticasone, consisting of 250μg fluticasone b.i.d for 6 weeks, followed by 100μg fluticasone b.i.d for 6 weeks, followed by placebo for 40 weeks (randomised treatment period).
Period: Overall Study
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Started | 1244 | 1244
Completed | 1016 (Includes open-label treatment if appropriate) | 1011 (Includes open-label treatment if appropriate)
Not Completed | 228 | 233
Not completed — Adverse Event | 108 | 101
Not completed — Lack of Efficacy | 6 | 6
Not completed — Protocol Violation | 27 | 23
Not completed — Lost to Follow-up | 9 | 7
Not completed — Withdrawal by Subject | 48 | 61
Not completed — Other reason not defined above | 29 | 33
Not completed — Not treated | 1 | 2

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) which included all patients who were dispensed study medication and were documented to have taken ≥1 dose of randomised treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal | Total
Number analyzed (Participants) | 1243 | 1242 | 2485
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.6) | 64.0 (8.4) | 63.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 230 | 206 | 436
  Male | 1013 | 1036 | 2049

OUTCOME MEASURES:

1. Primary Outcome: Time to First Moderate or Severe On-treatment COPD Exacerbation
Description: A Chronic Obstructive Pulmonary Disease (COPD) exacerbation was defined as an increase or new onset of ≥2 lower respiratory symptoms related to COPD, with ≥1 symptom lasting ≥3 days, requiring a change in treatment. Lower respiratory symptoms included shortness of breath, sputum production (volume), sputum purulence, cough, wheezing and chest tightness. A change in treatment included: hospitalisation/treatment in an urgent care unit, prescription of antibiotics and/or systemic steroids or a significant change of prescribed respiratory medication such as theophyllines, long-acting beta-agonists or inhaled corticosteroids. Exacerbations were considered severe if the patient was held and treated for an acute respiratory condition in an urgent care department or an observation unit for >6 hours, the patient was treated at home by a mobile urgent care team or the patient was admitted to hospital.The "measure type" displays the 25th percentile and its 95% confidence interval.
Time Frame: During randomised treatment, up to 488 days
Population: Treated set
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
days | 107.0 [94.0 to 124.0] | 110.0 [99.0 to 120.0]
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Test type: Non-Inferiority or Equivalence — Upper limit of 95% confidence interval (CI) <1.2 indicates non-inferiority of Fluticasone withdrawal compared with Fluticasone maintenance; p = 0.3497, Chi-squared — Two-sided p-value to test superiority of fluticasone maintenance over fluticasone withdrawal if non-inferiority shown; Wald's chi-square test; Hazard Ratio (HR) = 1.058, 95% CI 2-sided [0.941 to 1.189] — Ratio calculated as fluticasone withdrawal divided by fluticasone maintenance

2. Secondary Outcome: Number of Moderate or Severe On-treatment COPD Exacerbations
Description: Number of moderate or severe on-treatment COPD exacerbations, based on a 7-day gap rule: exacerbations where the onset date of the second exacerbation event was ≤7 days after the end date of the first exacerbation event were combined and counted as moderate or severe if ≥1 of the contributing exacerbation events was moderate or severe. Exacerbations were considered severe if the patient was held and treated for an acute respiratory condition in an urgent care department or an observation unit for >6 hours, the patient was treated at home by a mobile urgent care team or the patient was admitted to hospital. Exacerbations were considered moderate if they required prescription of antibiotics and/or systemic steroids.
  Measured values show adjusted mean event rate.
Time Frame: During randomised treatment, up to 488 days
Population: Treated Set
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient-year
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
exacerbations per patient-year | 0.91 [0.83 to 0.99] | 0.95 [0.87 to 1.04]
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Test type: Superiority or Other; p = 0.4441, Regression, Negative Binomial; Adjusted for log time at risk using log link function; Rate ratio = 1.05, 95% CI 2-sided [0.93 to 1.18], Standard Error of Mean 0.06 — Ratio calculated as fluticasone withdrawal divided by fluticasone maintenance

3. Secondary Outcome: Proportion of Patients With ≥1 Moderate or Severe On-treatment COPD Exacerbation
Description: Presence (yes vs no) of at least one moderate or severe on-treatment COPD exacerbation, displayed as a percentage. Exacerbations were considered severe if the patient was held and treated for an acute respiratory condition in an urgent care department or an observation unit for >6 hours, the patient was treated at home by a mobile urgent care team or the patient was admitted to hospital. Exacerbations were considered moderate if they required prescription of antibiotics and/or systemic steroids.
Time Frame: During randomised treatment, up to 488 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
percentage of participants | 44.2 | 46.7
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Test type: Superiority or Other; p = 0.2269, Fisher Exact

4. Secondary Outcome: Time to First Severe On-treatment COPD Exacerbation
Description: Time to first severe on-treatment COPD exacerbation. Exacerbations were considered severe if the patient was held and treated for an acute respiratory condition in an urgent care department or an observation unit for >6 hours, the patient was treated at home by a mobile urgent care team or the patient was admitted to hospital.
  The "measure type" displays the 25th percentile and its 95% confidence interval.
Time Frame: During randomised treatment, up to 488 days
Population: Treated set
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
days | NA [NA to NA] — Not estimable as not enough events during the timeframe. | 419.0 [379.0 to NA] — Not estimable as not enough events during the timeframe.
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Test type: Superiority or Other; p = 0.0849, Chi-squared; Wald's chi-square test; Hazard Ratio (HR) = 1.202, 95% CI 2-sided [0.975 to 1.481] — Ratio calculated as fluticasone withdrawal divided by fluticasone maintenance

5. Secondary Outcome: Number of Severe On-treatment COPD Exacerbations
Description: Number of severe on-treatment COPD exacerbations based on a 7-day gap rule: exacerbations where the onset date of the second exacerbation event was ≤7 days after the end date of the first exacerbation event were combined and counted as severe if ≥1 of the contributing exacerbation events was severe. Exacerbations were considered severe if the patient was held and treated for an acute respiratory condition in an urgent care department or an observation unit for >6 hours, the patient was treated at home by a mobile urgent care team or the patient was admitted to hospital.
  Measured values show adjusted event rate.
Time Frame: During randomised treatment, up to 488 days
Population: Treated set
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient-year
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
exacerbations per patient-year | 0.20 [0.17 to 0.23] | 0.23 [0.19 to 0.27]
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Test type: Superiority or Other; p = 0.2291, Regression, Negative Binomial; Adjusted for log time at risk using log link function; Rate ratio = 1.15, 95% CI 2-sided [0.92 to 1.45], Standard Error of Mean 0.13 — Ratio calculated as fluticasone withdrawal divided by fluticasone maintenance

6. Secondary Outcome: Proportion of Patients With at Least One Severe On-treatment COPD Exacerbation.
Description: Presence (yes vs no) of at least one severe on-treatment COPD exacerbation, displayed as a percentage. Exacerbations were considered severe if the patient was held and treated for an acute respiratory condition in an urgent care department or an observation unit for >6 hours, the patient was treated at home by a mobile urgent care team or the patient was admitted to hospital.
Time Frame: During randomised treatment, up to 488 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
percentage of participants | 13.4 | 15.2
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Test type: Superiority or Other; p = 0.2083, Fisher Exact

7. Secondary Outcome: Time to First On-treatment COPD Exacerbation
Description: Time to first on-treatment COPD exacerbation of any severity. The "measure type" displays the 25th percentile and its 95% confidence interval.
Time Frame: During randomised treatment, up to 488 days
Population: Treated set
Measure: Number (95% Confidence Interval); unit: days
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
days | 365.0 [309.0 to NA] — Not estimable as not enough events during the timeframe. | 346.0 [302.0 to NA] — Not estimable as not enough events during the timeframe.
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Test type: Superiority or Other; p = 0.5562, Chi-squared; Hazard Ratio (HR) = 1.035, 95% CI 2-sided [0.923 to 1.160]

8. Secondary Outcome: Number of On-treatment COPD Exacerbations
Description: Number of on-treatment COPD exacerbations of any severity, based on a 7-day gap rule: exacerbations where the onset date of the second exacerbation event was ≤7 days after the end date of the first exacerbation event were combined.
  Measured values show adjusted event rate.
Time Frame: During randomised treatment, up to 488 days
Population: Treated set
Measure: Mean (95% Confidence Interval); unit: exacerbations per patient-year
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
exacerbations per patient-year | 1.03 [0.95 to 1.12] | 1.08 [0.99 to 1.17]
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Test type: Superiority or Other; p = 0.4342, Regression, Negative binomial; Adjusted for log time at risk using log link function; Rate ratio = 1.05, 95% CI 2-sided [0.93 to 1.18], Standard Error of Mean 0.06 — Ratio calculated as fluticasone withdrawal divided by fluticasone maintenance

9. Secondary Outcome: Proportion of Patients With at Least One On-treatment COPD Exacerbation
Description: Presence (yes vs no) of at least one on-treatment COPD exacerbation of any severity, displayed as a percentage.
Time Frame: During randomised treatment, up to 488 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
percentage of participants | 46.9 | 49.0
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Test type: Superiority or Other; p = 0.3155, Fisher Exact

10. Secondary Outcome: Severity of On-treatment COPD Exacerbations
Description: Severity of on-treatment COPD exacerbations: for each patient, the worst applicable category was taken (i.e. none, mild, moderate or severe)
Time Frame: During randomised treatment, up to 488 days
Population: Treated set
Measure: Number; unit: percentage of participants
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
percentage of participants
  None and patient completed randomised treatment | 42.9 | 41.2
  None and patient discontinued randomised treatment | 10.2 | 9.8
  Mild | 2.7 | 2.3
  Moderate | 30.8 | 31.5
  Severe | 13.4 | 15.2

11. Secondary Outcome: Change in On-treatment Lung Function as Measured by Trough FEV1
Description: Change from baseline in on-treatment lung function as measured by trough forced expiratory volume in one second (FEV1); change was calculated as week score minus baseline score. Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 6, 12, 18 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
Litres
  Week 6 visit (N=1135, 1135) | -0.009 (0.0062) | -0.011 (0.0062)
  Week 12 visit (N=1114, 1092) | -0.011 (0.0062) | -0.018 (0.0063)
  Week 18 visit (N=1077, 1058) | -0.011 (0.0064) | -0.050 (0.0064)
  Week 52 visit (N=970, 935) | -0.016 (0.0094) | -0.059 (0.0096)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.0014, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = -0.043, 95% CI 2-sided [-0.069 to -0.017], Standard Error of Mean 0.0134 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

12. Secondary Outcome: Changes in On-treatment Dyspnoea as Measured by the Modified Medical Research Council (MMRC) Dyspnoea Scale
Description: Change from baseline in on-treatment dyspnoea as measured by the Modified Medical Research Council (MMRC) dyspnoea scale; change was calculated as week score minus baseline score. Negative changes from baseline indicate an improvement in health.
  Scale from 0 to 4:
  * 0 = not troubled by breathlessness, except during strenuous exercise
  * 1 = short of breath when hurrying or walking up a slight hill
  * 2 = walks slower than contemporaries on the same level because of breathlessness, or has to stop for breath when walking at own pace
  * 3 = stops for breath after approximately 100 yards, or after a few minutes on the level
  * 4 = too breathless to leave the house, or breathless when dressing or undressing
  "No breathlessness" was given a score of -1
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 18 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
units on a scale
  Week 18 visit (N=1140, 1143) | -0.030 (0.022) | -0.001 (0.022)
  Week 52 visit (N=1043, 1019) | -0.028 (0.024) | 0.035 (0.024)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.0632, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = 0.064, 95% CI 2-sided [-0.004 to 0.131], Standard Error of Mean 0.034 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

13. Secondary Outcome: Change in On-treatment Physical Health Status as Determined by Body Mass Index (BMI)
Description: Change from baseline in on-treatment physical health status as determined by body mass index (BMI); change was calculated as week score minus baseline score. Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 18 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: kg/m2
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
kg/m2
  Week 18 visit (N=1143, 1146) | 0.030 (0.028) | 0.040 (0.028)
  Week 52 visit (N=1047, 1021) | 0.004 (0.039) | -0.009 (0.039)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.8137, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = -0.013, 95% CI 2-sided [-0.122 to 0.096], Standard Error of Mean 0.055 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

14. Secondary Outcome: Change in On-treatment Exercise Capacity Measured by Six-minute Walk Test (6-MWT)
Description: Change from baseline in on-treatment exercise capacity measured by six-minute walk test (6-MWT); change was calculated as week score minus baseline score. Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 18 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
meters
  Week 18 visit (N=1111, 1110) | 3.89 (1.993) | 1.94 (1.993)
  Week 52 visit (N=1013, 987) | 3.94 (2.231) | 0.42 (2.252)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.2663, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = -3.53, 95% CI 2-sided [-9.74 to 2.69], Standard Error of Mean 3.170 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

15. Secondary Outcome: Change in On-treatment BODE Index
Description: Change from baseline in on-treatment BODE index (Body mass index, airflow Obstruction, Dyspnea and Exercise capacity index), a composite score ranging from 0 (best) to 10 (worst); change was calculated as week score minus baseline score. Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 18 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
units on a scale
  Week 18 visit (N=1038, 1024) | -0.06 (0.03) | 0.06 (0.03)
  Week 52 visit (N=931, 907) | -0.03 (0.04) | 0.14 (0.04)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.0033, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = 0.16, 95% CI 2-sided [0.05 to 0.27], Standard Error of Mean 0.06 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

16. Secondary Outcome: Change in On-treatment Cough and Expectoration as Measured by the CASA-Q: Cough Impact Domain
Description: Change from baseline in on-treatment cough and expectoration as measured by the cough and sputum assessment questionnaire (CASA-Q) (selected sites only): Cough impact domain. Change was calculated as week score minus baseline score. Response options for the items in this domain range from "not at all/never" to "extremely/always" on a five-point scale. Domain items were reverse scored, summed and transformed to a domain score ranging from 0 to 100 where a higher score is associated with less impact due to cough.
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 12, 18 and 52 visits
Population: Treated set who completed CASA-Q
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 364 | 361
units on a scale
  Week 12 visit (N=307, 319) | -1.65 (0.986) | -1.24 (0.968)
  Week 18 visit (N=302, 312) | -2.87 (1.035) | -3.71 (1.018)
  Week 52 visit (N=268, 269) | -4.51 (1.063) | -5.54 (1.057)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.4914, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = -1.03, 95% CI 2-sided [-3.98 to 1.91], Standard Error of Mean 1.499 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

17. Secondary Outcome: Change in On-treatment Cough and Expectoration as Measured by the CASA-Q: Cough Symptoms Domain
Description: Change from baseline in on-treatment cough and expectoration as measured by the cough and sputum assessment questionnaire (CASA-Q) (selected sites only): Cough symptoms domain. Change was calculated as week score minus baseline score. Response options for the items in this domain range from "not at all/never" to "a lot/always" on a five-point scale. Domain items were reverse scored, summed and transformed to a domain score ranging from 0 to 100 where a higher score is associated with less symptoms due to cough.
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 12, 18 and 52 visits
Population: Treated set who completed CASA-Q
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 364 | 361
units on a scale
  Week 12 visit (N=309, 318) | -0.32 (1.062) | -0.85 (1.048)
  Week 18 visit (N=305, 312) | -1.47 (1.103) | -3.34 (1.091)
  Week 52 visit (N=270, 268) | -1.69 (1.180) | -3.26 (1.180)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.3490, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = -1.56, 95% CI 2-sided [-4.84 to 1.71], Standard Error of Mean 1.669 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

18. Secondary Outcome: Change in On-treatment Cough and Expectoration as Measured by the CASA-Q: Sputum Impact Domain
Description: Change from baseline in on-treatment cough and expectoration as measured by the cough and sputum assessment questionnaire (CASA-Q) (selected sites only): Sputum impact domain. Change was calculated as week score minus baseline score. Response options for the items in this domain range from "not at all/never" to "a lot/always" on a five-point scale. Domain items were reverse scored, summed and transformed to a domain score ranging from 0 to 100 where a higher score is associated with less impact due to sputum.
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 12, 18 and 52 visits
Population: Treated set who completed CASA-Q
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 364 | 361
units on a scale
  Week 12 visit (N=308, 317) | -2.26 (0.996) | -1.63 (0.983)
  Week 18 visit (N=303, 310) | -2.38 (0.977) | -3.31 (0.967)
  Week 52 visit (N=267, 267) | -4.29 (1.047) | -4.15 (1.045)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.9262, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = 0.14, 95% CI 2-sided [-2.77 to 3.04], Standard Error of Mean 1.480 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

19. Secondary Outcome: Change in On-treatment Cough and Expectoration as Measured by the CASA-Q: Sputum Symptoms Domain
Description: Change from baseline in on-treatment cough and expectoration as measured by the cough and sputum assessment questionnaire (CASA-Q) (selected sites only): Sputum symptoms domain. Change was calculated as week score minus baseline score. Response options for the items in this domain range from "not at all/never" to "extremely/always" on a five-point scale. Domain items were reverse scored, summed and transformed to a domain score ranging from 0 to 100 where a higher score is associated with less symptoms due to sputum.
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 12, 18 and 52 visits
Population: Treated set who completed CASA-Q
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 364 | 361
units on a scale
  Week 12 visit (N=308, 317) | -1.36 (1.154) | -1.24 (1.139)
  Week 18 visit (N=302, 311) | -2.71 (1.119) | -1.93 (1.105)
  Week 52 visit (N=269, 268) | -5.10 (1.212) | -2.45 (1.211)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.1241, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = 2.64, 95% CI 2-sided [-0.73 to 6.01], Standard Error of Mean 1.716 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

20. Secondary Outcome: Change in On-treatment FEV1 as Measured by Home Based Spirometry
Description: Change from baseline in on-treatment Forced Expiratory Volume in One Second (FEV1) as measured by home based spirometry. Change was calculated as week score minus baseline score. The weekly mean was defined as the mean of the measurements taken during the last 7 days prior to the visit date, and was calculated if ≥4 of the 7 days had non-missing measurements. Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 6, 12, 18, 27, 36, 45 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
Litres
  Week 6 visit (N=893, 939) | -0.049 (0.0066) | -0.053 (0.0065)
  Week 12 visit (N=910, 930) | -0.050 (0.0068) | -0.056 (0.0067)
  Week 18 visit (N=913, 901) | -0.051 (0.0068) | -0.093 (0.0068)
  Week 27 visit (N=863, 843) | -0.056 (0.0071) | -0.092 (0.0072)
  Week 36 visit (N=854, 845) | -0.059 (0.0074) | -0.099 (0.0074)
  Week 45 visit (N=830, 815) | -0.061 (0.0080) | -0.103 (0.0080)
  Week 52 visit (N=785, 788) | -0.067 (0.0087) | -0.115 (0.0087)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p < 0.0001, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = -0.048, 95% CI 2-sided [-0.073 to -0.024], Standard Error of Mean 0.0123 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

21. Secondary Outcome: Change in On-treatment FVC as Measured by Home Based Spirometry
Description: Change from baseline in on-treatment forced vital capacity (FVC) as measured by home based spirometry. Change was calculated as week score minus baseline score. The weekly mean was defined as the mean of the measurements taken during the last 7 days prior to the visit date, and was calculated if ≥4 of the 7 days had non-missing measurements. Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 6, 12, 18, 27, 36, 45 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
Litres
  Week 6 visit (N=893, 939) | -0.116 (0.0179) | -0.089 (0.0177)
  Week 12 visit (N=910, 930) | -0.113 (0.0168) | -0.105 (0.0167)
  Week 18 visit (N=913, 901) | -0.122 (0.0177) | -0.124 (0.0177)
  Week 27 visit (N=863, 843) | -0.123 (0.0167) | -0.147 (0.0167)
  Week 36 visit (N=854, 845) | -0.135 (0.0170) | -0.158 (0.0171)
  Week 45 visit (N=830, 815) | -0.141 (0.0174) | -0.168 (0.0175)
  Week 52 visit (N=785, 788) | -0.157 (0.0180) | -0.201 (0.0180)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.0855, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = -0.044, 95% CI 2-sided [-0.094 to 0.006], Standard Error of Mean 0.0255 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

22. Secondary Outcome: Change in On-treatment PEFR as Measured by Home Based Spirometry
Description: Change from baseline in on-treatment peak expiratory flow rate (PEFR) as measured by home based spirometry; change was calculated as week score minus baseline score. Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 6, 12, 18, 27, 36, 45 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: Litres/sec
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
Litres/sec
  Week 6 visit (N=893, 939) | -0.228 (0.0249) | -0.230 (0.0246)
  Week 12 visit (N=910, 930) | -0.266 (0.0253) | -0.290 (0.0252)
  Week 18 visit (N=913, 901) | -0.295 (0.0253) | -0.435 (0.0254)
  Week 27 visit (N=863, 843) | -0.319 (0.0273) | -0.430 (0.0274)
  Week 36 visit (N=854, 845) | -0.352 (0.0278) | -0.473 (0.0278)
  Week 45 visit (N=830, 815) | -0.368 (0.0297) | -0.490 (0.0298)
  Week 52 visit (N=785, 788) | -0.377 (0.0318) | -0.538 (0.0318)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.0004, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = -0.161, 95% CI 2-sided [-0.249 to -0.073], Standard Error of Mean 0.0450 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

23. Secondary Outcome: Change in On-treatment St Georges Respiratory Questionnaire (SGRQ) Scores: Activity Domain
Description: Change from baseline in on-treatment St Georges Respiratory Questionnaire (SGRQ) scores: Activity domain. Scores range from 0 to 100, with higher scores indicating more limitations. Change was calculated as week score minus baseline score.
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 27 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
units on a scale
  Week 27 visit (N=1002, 988) | 0.09 (0.492) | 0.85 (0.496)
  Week 52 visit (N=942, 916) | -0.19 (0.512) | 0.78 (0.518)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.1838, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = 0.97, 95% CI 2-sided [-0.46 to 2.40], Standard Error of Mean 0.728 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

24. Secondary Outcome: Change in On-treatment St Georges Respiratory Questionnaire (SGRQ) Scores: Impact Domain
Description: Change from baseline in on-treatment St Georges Respiratory Questionnaire (SGRQ) scores: Impact Domain. Scores range from 0 to 100, with higher scores indicating more limitations. Change was calculated as week score minus baseline score.
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 27 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
units on a scale
  Week 27 visit (N=1004, 998) | -0.78 (0.456) | 0.35 (0.457)
  Week 52 visit (N=946, 921) | -0.08 (0.494) | 1.27 (0.499)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.0551, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = 1.35, 95% CI 2-sided [-0.03 to 2.72], Standard Error of Mean 0.702 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

25. Secondary Outcome: Change in On-treatment St Georges Respiratory Questionnaire (SGRQ) Scores: Symptoms Domain
Description: Change from baseline in on-treatment St Georges Respiratory Questionnaire (SGRQ) scores: Symptoms domain. Scores range from 0 to 100, with higher scores indicating more limitations. Change was calculated as week score minus baseline score.
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 27 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
units on a scale
  Week 27 visit (N=1010, 998) | 0.12 (0.583) | 0.62 (0.586)
  Week 52 visit (N=955, 921) | 0.51 (0.593) | 1.11 (0.602)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.4804, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = 0.60, 95% CI 2-sided [-1.06 to 2.25], Standard Error of Mean 0.845 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

26. Secondary Outcome: Change in On-treatment St Georges Respiratory Questionnaire (SGRQ) Scores: Total Score
Description: Change from baseline in on-treatment St Georges Respiratory Questionnaire (SGRQ) scores: Total score. Scores range from 0 to 100, with higher scores indicating more limitations. Change was calculated as week score minus baseline score.
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 27 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
units on a scale
  Week 27 visit (N=996, 986) | -0.42 (0.398) | 0.55 (0.401)
  Week 52 visit (N=939, 913) | -0.07 (0.432) | 1.15 (0.437)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.0467, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = 1.22, 95% CI 2-sided [0.02 to 2.43], Standard Error of Mean 0.614 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

27. Secondary Outcome: Change in On-treatment Physician Global Evaluation
Description: Change from baseline in on-treatment physician global evaluation. The evaluation reflected the physician's opinion of the patient's overall condition and was based on the need for concomitant medication, the number and severity of exacerbations, the severity of cough, the ability to exercise, the amount of wheezing and any other relevant clinical observations. Patients were graded on a scale of 1 (poor) to 8 (excellent). Change was calculated as week score minus baseline score.
  Statistical analysis results are presented only for the week 52 visit as this is the primary timepoint of interest.
Time Frame: Baseline and week 27 and 52 visits
Population: Treated set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Number analyzed (Participants) | 1243 | 1242
units on a scale
  Week 27 visit (N=1113, 1093) | 0.10 (0.03) | 0.04 (0.03)
  Week 52 visit (N=1041, 1014) | 0.19 (0.03) | 0.08 (0.03)
Statistical Analysis 1: Comparison: Fluticasone Maintenance vs Fluticasone Withdrawal; Week 52 visit; Test type: Superiority or Other; p = 0.0223, Restricted maximum likelihood; Repeated measures restricted maximum likelihood; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.21 to -0.02], Standard Error of Mean 0.05 — Difference calculated as fluticasone withdrawal minus fluticasone maintenance

ADVERSE EVENTS:
Time Frame: Randomised treatment plus 30 days post-treatment for patients not switching to open-label, up to 518 days
Arm/Group | Fluticasone Maintenance | Fluticasone Withdrawal
Serious Adverse Events (participants affected / at risk) | 292/1243 | 300/1242
Other Adverse Events (participants affected / at risk) | 464/1243 | 458/1242
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Maintenance (N=1243) | Fluticasone Withdrawal (N=1242)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 5 | 1
Angina pectoris (Cardiac disorders) | 2 | 1
Angina unstable (Cardiac disorders) | 4 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 3 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 9 | 5
Atrial flutter (Cardiac disorders) | 3 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 3 | 4
Cardiac asthma (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 3
Cardiac failure acute (Cardiac disorders) | 1 | 2
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Cor pulmonale (Cardiac disorders) | 2 | 2
Cor pulmonale chronic (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 1
Hypertensive heart disease (Cardiac disorders) | 1 | 2
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 2
Myocardial ischaemia (Cardiac disorders) | 4 | 0
Right ventricular failure (Cardiac disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 3 | 4
Pterygium (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colonic stenosis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Oesophageal food impaction (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 3
Death (General disorders) | 0 | 2
Impaired healing (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 3
Sudden death (General disorders) | 1 | 3
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 3
Bronchitis bacterial (Infections and infestations) | 0 | 2
Bronchopneumonia (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Escherichia infection (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 7 | 5
Klebsiella infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 12 | 3
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 1 | 2
Meningitis viral (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 34 | 38
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 3
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 2
Tracheobronchitis (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Vestibular neuronitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Bronchitis chemical (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Burns third degree (Injury, poisoning and procedural complications) | 1 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 2
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Scrotal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Urethral injury (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
Angiogram (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Pulmonary function test decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Maxillofacial sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Oropharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Vocal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 2
Cerebral microangiopathy (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 1
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 2
Intercostal neuralgia (Nervous system disorders) | 1 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Meningorrhagia (Nervous system disorders) | 0 | 1
Radiculitis cervical (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Renal failure chronic (Renal and urinary disorders) | 4 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Urethral haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 2 | 2
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bullous lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 154 | 180
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Laryngeal leukoplakia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Alcohol detoxification (Surgical and medical procedures) | 1 | 0
Angioplasty (Surgical and medical procedures) | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 0
Oxygen supplementation (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 1 | 0
Aortic aneurysm (Vascular disorders) | 2 | 1
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 2
Arteriosclerosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 3
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 2 | 0
Phlebitis (Vascular disorders) | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Maintenance (N=1243) | Fluticasone Withdrawal (N=1242)
Nasopharyngitis (Infections and infestations) | 93 | 80
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 410 | 413

LIMITATIONS AND CAVEATS:
Additional secondary endpoints were listed in the original protocol. Those endpoints are of exploratory nature only and were not considered relevant for trial conclusions. For more information see tab "Full Text Review", section "More Information".

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.